CLINICAL TRIAL: NCT07052331
Title: The MOBY Study - Efficacy of Birth Mobility: Randomized Clinical Trial Investigating the Efficacy of Birth Mobility on Birth Outcomes in Primiparous Women With and Without a Birth Mobility System.
Brief Title: The MOBY Study: Efficacy of Birth Mobility
Acronym: MOBY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vibwife AG (Industry)
Collaborators: Kantonsspital Baden (Other); Fachhochschule Nordwestschweiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-D0016; 103.215 IP-LS (Other Grant/Funding Number: INNOSUISSE); 2025-D0016 (Registry Identifier: Swiss National Clinical Trials Portal (SNCTP))
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Labor Duration; Cesarean Section Rate; Maternal Mobility; Healthy
Keywords: Birth mobility; Maternal satisfaction; Labor and delivery; Neonatal outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Birth Mobility System (Experimental): Participants receive standard obstetric care and have access to a birth mobility system installed on the birthing bed. Use of the system is voluntary and guided by medical professionals. Participants view a video explaining the system's operation. Birth mobility data is collected passively.
  Interventions: Device: Birth Mobility System
- Standard obstetric care (No Intervention): Participants receive standard obstetric care using a conventional birthing bed. No access is given to the birth mobility system. Birth mobility data is collected passively.

INTERVENTIONS:
Device: Birth Mobility System — Participants receive standard obstetric care and have access to a birth mobility system installed on the birthing bed. Use of the system is voluntary and guided by medical professionals. Participants view a video explaining the system's operation. Birth mobility data is collected passively.
  Arms: Birth Mobility System

SUMMARY:
This randomized clinical trial investigates whether and how maternal mobility during labor influences birth outcomes in primiparous women. The study compares standard obstetric care with care that includes a birth mobility system. The primary aim is to assess whether the system helps reduce secondary cesarean section rates. Secondary objectives include evaluation of labor progression, medication use, newborn health, and user satisfaction. Participation occurs during birth and includes the collection of routine clinical data and a short questionnaire afterward.

DETAILED DESCRIPTION:
The MOBY study is a randomized clinical investigation evaluating the efficacy of maternal birth mobility on delivery outcomes in first-time mothers. The study takes place at Kantonsspital Baden and includes 714 participants.

The aim of the study is to examine whether certain positions and mobility during labor can positively influence the birth process. These insights may improve support for women in labor in the future.

Participants are randomly assigned to one of two groups:

The control group receives the usual hospital infrastructure, including a conventional static birthing bed.

The intervention group receives, in addition to standard care, access to a CE-marked birth mobility system that offers supportive movement options. Participants in this group are shown a short instructional video.

In both groups, positioning and movement during labor are recorded passively using a non-intrusive monitoring setup. These recordings are not noticeable for the participants and do not interfere with clinical care. The medical team continues to provide position recommendations according to each individual situation and based on current standards in midwifery and obstetrics. Women are always free to move and position themselves as they wish.

After birth, participants are asked to complete a short questionnaire about their birth experience. A similar questionnaire is completed by the midwife.

The primary objective is to determine whether the use of the birth mobility system is associated with a lower rate of secondary cesarean sections. Secondary objectives include analysis of labor duration, analgesia and oxytocin use, pain levels, birth mode, neonatal outcomes, and satisfaction of participants and healthcare providers. In addition, movement characteristics observed during labor will be explored to support future research and care improvements.

This is a Category A1 study involving CE-marked medical devices used according to their intended purpose. The study follows ISO 14155, the current version of the Declaration of Helsinki, ICH-GCP, and all legally applicable national regulations. The study has been approved by the responsible Ethics Committee (EKNZ). All personal data are pseudonymized and handled in compliance with Swiss and international data protection standards. No risks beyond standard obstetric care are introduced by participation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* German- or English-speaking
* Able to provide written informed consent with capacity of judgment
* Low-risk singleton pregnancy
* Primiparous woman
* Cephalic presentation
* Gestational age at delivery ≥ 37 + 0 weeks

Exclusion Criteria:

* Multiparous woman
* Not capable of understanding instructions for use of the mobility system (intervention group)
* Scheduled (elective) cesarean section
* Contraindication to vaginal delivery
* Multiple pregnancy
* Breech presentation
* Estimated fetal weight < 10th percentile or > 90th percentile
* Relevant fetal congenital abnormalities affecting neonatal adaptation
* Pre-existing medical conditions significantly affecting mobility (e.g., orthopedic conditions, osteoporosis, multiple sclerosis, spinal cord injury)
* Relevant intrapartum bleeding
* Preeclampsia or HELLP syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Rate of Secondary Cesarean Section | At birth
  The proportion of women who undergo a cesarean section after the onset of labor (i.e. unplanned cesarean section).

SECONDARY OUTCOMES:
Mode of Delivery | At birth
  Categorized as vaginal, vaginal-operative, or cesarean section, based on hospital documentation.
Duration of Labor | From clinical onset of first stage of labor (regular contractions with cervical dilation > 3-4cm) until birth.
  Measured separately for the first and second stages of labor in minutes.
Use of Epidural Anesthesia | During labor
  Binary outcome (yes/no), recorded from medical records.
Use of Opioid Analgesia | During labor
  Binary outcome (yes/no), recorded from hospital medication records.
Use of Oxytocin During Labor | During labor
  Binary outcome (yes/no), recorded from clinical records.
Maternal Pain Score (NRS) | During labor until immediately after birth
  Numeric Rating Scale (0-10) reported by the participant to quantify perceived pain during labor.
Umbilical Artery pH Value | Immediately after birth
  Value measured from cord blood sample at birth to assess fetal oxygenation.
APGAR Score at 10 Minutes | 10 minutes after birth
  Standardized score (0-10) assessing newborn health at 10 minutes after delivery.
Maternal Satisfaction With Birth Experience | Within 2 hours after birth
  Measured via a post-birth questionnaire completed by the participant (Likert-type scale).
Healthcare Professional Satisfaction | Within 2 hours after birth
  Measured using a structured questionnaire completed by the attending midwife after each birth.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Leonhard Schäffer, Principal Investigator — Kantonsspital Baden
Locations (1):
- Kantonsspital Baden, Baden, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared in order to fully protect participant privacy. Although the data are pseudonymized, elements such as birth date and detailed clinical information in a single-site population may still carry a risk of re-identification. In accordance with Swiss data protection law and ethics approval conditions, only aggregated and anonymized results will be published.

REFERENCES:
- [Background] Opiyo N, Kingdon C, Oladapo OT, Souza JP, Vogel JP, Bonet M, Bucagu M, Portela A, McConville F, Downe S, Gulmezoglu AM, Betran AP. Non-clinical interventions to reduce unnecessary caesarean sections: WHO recommendations. Bull World Health Organ. 2020 Jan 1;98(1):66-68. doi: 10.2471/BLT.19.236729. Epub 2019 Nov 29. No abstract available. PMID 31902964
- [Background] Romano AM, Lothian JA. Promoting, protecting, and supporting normal birth: a look at the evidence. J Obstet Gynecol Neonatal Nurs. 2008 Jan-Feb;37(1):94-104; quiz 104-5. doi: 10.1111/j.1552-6909.2007.00210.x. PMID 18226163
- [Background] Hanson L. Second-stage labor care: challenges in spontaneous bearing down. J Perinat Neonatal Nurs. 2009 Jan-Mar;23(1):31-9; quiz 40-1. doi: 10.1097/JPN.0b013e318196526b. PMID 19209057
- [Background] Monod C, Granado C, Mueller D, Gisin M, Ries JJ, Horn S, Erlanger TE, Hoesli I. Safety and acceptance of "Vibwife", a new moving mattress to support mobilization during labor: Result of a clinical study. Midwifery. 2021 Dec;103:103096. doi: 10.1016/j.midw.2021.103096. Epub 2021 Jul 17. PMID 34311336
- [Background] Ondeck M. Healthy birth practice #2: walk, move around, and change positions throughout labor. J Perinat Educ. 2014 Fall;23(4):188-93. doi: 10.1891/1058-1243.23.4.188. PMID 25411538
- [Background] Roberts J, Hanson L. Best practices in second stage labor care: maternal bearing down and positioning. J Midwifery Womens Health. 2007 May-Jun;52(3):238-45. doi: 10.1016/j.jmwh.2006.12.011. PMID 17467590
- [Background] Lawrence A, Lewis L, Hofmeyr GJ, Styles C. Maternal positions and mobility during first stage labour. Cochrane Database Syst Rev. 2013 Aug 20;(8):CD003934. doi: 10.1002/14651858.CD003934.pub3. PMID 23959763